CLINICAL TRIAL: NCT00524680
Title: Study of Serum 25(OH) D3 Level Variability in Response to Different Doses of Oral Vitamin D Supplementation in Prostate Cancer Patients
Brief Title: Vitamin D in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000562742; I 95406 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive 4,000 IU of oral cholecalciferol (vitamin D3) once daily.
  Interventions: Dietary Supplement: cholecalciferol
- Arm II (Experimental): Patients receive 6,000 IU of vitamin D3 once daily.
  Interventions: Dietary Supplement: cholecalciferol
- Arm III (Experimental): Patients receive 8,000 IU of vitamin D3 once daily.
  Interventions: Dietary Supplement: cholecalciferol
- Arm IV (Experimental): Patients receive 10,000 IU of vitamin D3 once daily.
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given orally

SUMMARY:
RATIONALE: Vitamin D may be effective in treating patients with prostate cancer.

PURPOSE: This randomized phase II trial is studying how well 4 different doses of vitamin D works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine the pattern of response of serum 25(OH) D3 levels following cholecalciferol (vitamin D3) supplementation at four different oral doses in patients with prostate cancer.

Secondary

* To examine the pattern of response of parathormone (PTH) following vitamin D3 supplementation in these patients.
* To assess the toxicity of vitamin D3 supplementation in men with prostate cancer.

Tertiary

* To track occurrence of infections, deep vein thrombosis, vascular events, and falls in these patients.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive 4,000 IU of oral cholecalciferol (vitamin D3) once daily.
* Arm II: Patients receive 6,000 IU of vitamin D3 once daily.
* Arm III: Patients receive 8,000 IU of vitamin D3 once daily.
* Arm IV: Patients receive 10,000 IU of vitamin D3 once daily. Treatment in all arms continues for 6 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* 25(OH) D3 level < 80 ng/mL

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL
* Corrected serum calcium ≤ 10.5 mg/dL

Exclusion criteria:

* History of malabsorption syndrome (e.g., pancreatic insufficiency, celiac disease, or tropical sprue)
* Hypersensitivity to cholecalciferol or one of its components

PRIOR CONCURRENT THERAPY:

* No other concurrent vitamin D supplementation

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 148 patients were treated but only 128 patients were eligible for study outcome analysis.
Groups:
- Arm I: Vitamin D 4000 IU Daily: Patients receive 4,000 IU of oral cholecalciferol (vitamin D3) once daily.
  cholecalciferol: Given orally
- Arm II: Vitamin D 6000 IU Daily: Patients receive 6,000 IU of vitamin D3 once daily.
  cholecalciferol: Given orally
- Arm III: Vitamin D 8000 IU Daily: Patients receive 8,000 IU of vitamin D3 once daily.
  cholecalciferol: Given orally
- Arm IV: Vitamin D 10,000 IU Daily: Patients receive 10,000 IU of vitamin D3 once daily.
  cholecalciferol: Given orally
Period: Overall Study
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Started | 37 | 35 | 36 | 40
Completed | 34 | 34 | 33 | 34
Not Completed | 3 | 1 | 3 | 6
Not completed — progression | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily | Total
Number analyzed (Participants) | 37 | 35 | 36 | 40 | 148
Age, Continuous [Median (Standard Deviation); unit: years] | 68.2 (8.1) | 65.4 (8.7) | 67.9 (8.7) | 66.4 (9.3) | 66.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 37 | 35 | 36 | 40 | 148

OUTCOME MEASURES:

1. Primary Outcome: Pattern of Response of Serum 25(OH) D3 Levels
Description: Change from Baseline in Serum 25(OH) D3 Levels at 1, 3, and 6 Months at dose levels 4000, 6000, 8000 and 10000 IU. Statistical analysis was done using one sample t-test.
Time Frame: Baseline, at 1, 3, 6 months
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Number analyzed (Participants) | 33 | 31 | 32 | 32
ng/mL
  1-month | 11.34 (13.03) | 24.84 (16.18) | 18.87 (22.25) | 26.91 (16.1)
  3-month | 23.45 (11.99) | 38.31 (22.24) | 35.76 (26.28) | 45.67 (21.5)
  6-month | 27.16 (15.69) | 43.4 (29.28) | 41.7 (27.07) | 57.59 (27.91)
Statistical Analysis 1: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 1-Month for dose level 4000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 3-Month for dose level 4000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 6-Month for dose level 4000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 1-Month for dose level 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 3-Month for dose level 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 6-Month for dose level 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 1-Month for dose level 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 3-Month for dose level 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 9: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 6-Month for dose level 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 10: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 1-Month for dose level 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 11: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 3-Month for dose level 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 12: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in Serum 25(OH) D3 Levels at 6-Month for dose level 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < .0001, t-test, 2 sided

2. Secondary Outcome: Pattern of Response of Parathormone
Description: Change from Baseline in PTH Levels at 1, 3, and 6 Months at dose levels 4000, 6000, 8000 and 10000 IU. Statistical analysis was done using one sample t-test.
Time Frame: Baseline, at 1, 3, 6 months
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Number analyzed (Participants) | 33 | 31 | 32 | 32
pg/mL
  1-month | -.73 (18.82) | -12.18 (43.33) | -1.28 (31.84) | -10.37 (46.24)
  3-month | -11.3 (37.99) | .24 (34.01) | -8.03 (32.77) | -18.06 (35.31)
  6-month | -8.4 (33.05) | -24.05 (26.77) | -9.78 (34.22) | -16.51 (45.94)
Statistical Analysis 1: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in PTH Levels at 1-month for 4000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.8244, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in PTH Levels at 3-month for 4000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.1025, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm I: Vitamin D 4000 IU Daily; Change from Baseline in PTH Levels at 6-Month for dose level 4000 IU; Test type: Superiority or Other; p = 0.1744, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in PTH Levels at 1-month for 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.1281, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in PTH Levels at 3-month for 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.9688, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm II: Vitamin D 6000 IU Daily; Change from Baseline in PTH Levels at 6-month for 6000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in PTH Levels at 1-month for 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.8241, t-test, 2 sided
Statistical Analysis 8: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in PTH Levels at 3-month for 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.1828, t-test, 2 sided
Statistical Analysis 9: Comparison: Arm III: Vitamin D 8000 IU Daily; Change from Baseline in PTH Levels at 6-month for 8000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.1348, t-test, 2 sided
Statistical Analysis 10: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in PTH Levels at 1-month for 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.2214, t-test, 2 sided
Statistical Analysis 11: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in PTH Levels at 3-month for 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.0079, t-test, 2 sided
Statistical Analysis 12: Comparison: Arm IV: Vitamin D 10,000 IU Daily; Change from Baseline in PTH Levels at 6-month for 10000 IU. Statistical analysis was done using one sample t-test; Test type: Superiority or Other; p = 0.0631, t-test, 2 sided

3. Secondary Outcome: Toxicity
Description: Number of treated patients that had serious adverse events.
Time Frame: Baseline, at 1, 3 and 6 months
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Number analyzed (Participants) | 37 | 35 | 36 | 40
participants | 2 | 0 | 1 | 5

4. Secondary Outcome: Occurrence of Infections, Deep Vein Thrombosis, Vascular Events, and Falls
Description: Number of participant with occurrence of infections, deep venous thrombosis, vascular events and falls
Time Frame: Baseline, at 1, 3 ,6 months
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Number analyzed (Participants) | 37 | 35 | 36 | 40
participants | 2 | 0 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Arm I: Vitamin D 4000 IU Daily | Arm II: Vitamin D 6000 IU Daily | Arm III: Vitamin D 8000 IU Daily | Arm IV: Vitamin D 10,000 IU Daily
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/35 | 1/36 | 5/40
Other Adverse Events (participants affected / at risk) | 3/37 | 3/35 | 3/36 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Vitamin D 4000 IU Daily (N=37) | Arm II: Vitamin D 6000 IU Daily (N=35) | Arm III: Vitamin D 8000 IU Daily (N=36) | Arm IV: Vitamin D 10,000 IU Daily (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Radical prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Vitamin D 4000 IU Daily (N=37) | Arm II: Vitamin D 6000 IU Daily (N=35) | Arm III: Vitamin D 8000 IU Daily (N=36) | Arm IV: Vitamin D 10,000 IU Daily (N=40)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes